CLINICAL TRIAL: NCT00462813
Title: An Investigation Into the Effects of Diidolylmethane (BioResponse DIM®) Supplementation in Women With Low-Grade Cervical Cytological Abnormalities [CRISP-1]
Brief Title: Diindolylmethane in Treating Patients With Abnormal Cervical Cells
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barts and the London School of Medicine and Dentistry (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CRUK-CRISP-1; CDR0000539352 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN47437431; EU-20717
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2008-09

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3; cervical intraepithelial neoplasia grade 1
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Polymerase Chain Reaction; Vaginal Smears

INTERVENTIONS:
Drug: oral microencapsulated diindolylmethane
Genetic: polymerase chain reaction
Other: cervical Papanicolaou test
Other: cytology specimen collection procedure
Procedure: colposcopic biopsy

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of diindolylmethane, a substance found in cruciferous vegetables, may keep cervical intraepithelial neoplasia or cervical cancer from forming.

PURPOSE: This randomized phase III trial is studying diindolylmethane to see how well it works compared to a placebo in treating patients with abnormal cervical cells.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of diindolylmethane vs placebo in reducing the prevalence of histologically proven high-grade cervical intraepithelial neoplasia in patients with low-grade cervical cytological abnormalities.
* Compare the effect of these regimens in reducing the prevalence of cytological abnormalities in these patients.
* Compare the effect of these regimens in changing the clinical appearance of the cervix in these patients.
* Determine if diindolylmethane offers benefits in relation to human papillomavirus (HPV) status, including HPV type, viral load, and integration.
* Determine the side effects of supplementation with diindolylmethane.
* Determine the effects of this drug on migraine, mastalgia, weight, and premenstrual syndrome (PMS).

OUTLINE: This is a double-blind, randomized, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral diindolylmethane once daily for 6 months.
* Arm II: Patients receive oral placebo once daily for 6 months. Patients undergo cervical sampling at baseline and at 6 months for Pap testing by liquid based cytology and human papillomavirus (HPV) testing by polymerase chain reaction. Some patients also undergo urine and hair sample collection at baseline and at 3 and 6 months. Samples are analyzed for estrogen and diindolylmethane metabolites, to monitor patient compliance and response to treatment. Some patients have a cervical photograph taken using a colposcope at baseline and at 6 months. All patients undergo colposcopy at 6 months.

Patients complete a questionnaire at baseline (i.e., for reproductive history, diet, smoking, and premenstrual symptoms) and at 6 months (i.e., for side effects, compliance, changes in smoking, and contraception use). Patients with moderate to severe premenstrual syndrome (PMS) also complete PMS questionnaires once monthly during months 1-6 and 4 months following completion of study therapy. All patients are instructed to maintain current diet and to keep cruciferous vegetables and soy products constant during study course.

After completion of study treatment, patients are followed periodically for up to 7 years.

PROJECTED ACCRUAL: A total of 3,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* First mildly dyskaryotic Pap smear or a second borderline Pap smear taken within the Cervical Screening Wales program

  * Patients under surveillance following treatment for high-grade cervical intraepithelial neoplasia are not eligible
* No clinical suspicion of a concurrent invasive cervical cancer

PATIENT CHARACTERISTICS:

* No invasive cancer within the past 3 years
* No known HIV positivity
* Not pregnant or nursing
* Not planning to become pregnant within the next 6 months

PRIOR CONCURRENT THERAPY:

* No concurrent immunosuppressive drugs, warfarin, or theophylline
* No concurrent proton pump inhibitor drugs for ulcer or reflux disease (i.e., rabeprazole, esomeprazole magnesium, lansoprazole, omeprazole, or pantoprazole sodium)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Biopsy confirmed high-grade cervical intraepithelial neoplasia (CIN) at 6 months

SECONDARY OUTCOMES:
Change in lesion size at 6 months
Human papillomavirus (HPV) status and characteristics (type, viral load, and integration) at baseline and 6 months
Change in cervical cytology at 6 months
CIN ≥ grade 3 on histology at 6 months
Long term follow-up (i.e., 7 years)
Migraine, premenstrual syndrome (PMS), menstruation, and body weight

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sasieni, MD, Study Chair — Barts and the London School of Medicine and Dentistry
Locations (2):
- United Kingdom (2):
  - Barts and the London School of Medicine, London, England
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- See also: Effect of diindolylmethane supplementation on low-grade cervical cytological abnormalities: double-blind, randomised, controlled trial. Br J Cancer. 2012 Jan 3;106(1):45-52. doi: 10.1038/bjc.2011.496. Epub 2011 Nov 10. — http://www.ncbi.nlm.nih.gov/pubmed/22075942